CLINICAL TRIAL: NCT04129346
Title: Technology-Supported Physical Activity Intervention for Metastatic Breast Cancer Survivors: Fit2ThriveMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Siobhan M Phillips, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SP00049673; R21CA239130 (NIH)
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Breast Cancer; Obesity
Keywords: Inactivity; Breast Cancer; Metastatic Breast Cancer; Quality of life; Sedentary
MeSH Terms: conditions — Breast Neoplasms; Obesity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fit2ThriveMB (Experimental): Participants assigned to the Fit2ThriveMB will receive the Fit2ThriveMB smartphone app, Fitbit, and coaching calls.
  Interventions: Behavioral: Fit2ThriveMB App; Behavioral: Fitbit; Behavioral: Physical Activity Coaching Calls
- Healthy Living Control (Active Comparator): Participants in the healthy living group will receive the American Society of Cancer Oncologists smartphone app, cancer.net. They will also receive calls during the intervention period and the Fitbit following completion of 12 week assessments
  Interventions: Behavioral: Healthy Living Coaching Calls; Behavioral: Cancer.net app

INTERVENTIONS:
Behavioral: Fit2ThriveMB App — The Fit2thriveMB app will encourage participants to increase their physical activity. Participants will be provided with educational information on physical activity and effective behavior change strategies for incorporating more physical activity into their daily lives to increase their step count. Participants will be prompted each morning to report the intensity of their symptom burden (0 to 10). Based on their symptom rating and their previous day's step counts, participants will be provided with three different options or levels of goals for that day to either increase or decrease 10-20% or remain constant.
  Arms: Fit2ThriveMB
Behavioral: Fitbit — The Fitbit measures PA intensity, steps, and heart rate and syncs directly with the smartphone and will automatically sync with the Fit2ThriveMB app and provide Fitbit data to the study team in real-time.
  Arms: Fit2ThriveMB
Behavioral: Physical Activity Coaching Calls — Participants will receive weekly coaching calls which will: a) provide feedback on the previous week's symptom burden and progress on PA goals; b) review personalized goals and strategies for increasing PA for the next week; c) provide instruction on effective behavioral change techniques
  Arms: Fit2ThriveMB
Behavioral: Healthy Living Coaching Calls — Participants will receive weekly calls that will cover health and well-being topics for instance: symptom and stress management, healthy diet, hydration, sun safety, sleep hygiene, and meditation.
  Arms: Healthy Living Control
Behavioral: Cancer.net app — Cancer.net app content includes information about health and well-being, treatment guidelines specific to cancer type, symptom tracking and medication tracking
  Arms: Healthy Living Control

SUMMARY:
This study will test the feasibility and acceptability of increasing PA in metastatic breast cancer (MBC) patients using a smartphone app, fitbit and coaching.

DETAILED DESCRIPTION:
The primary purpose of the present study is to pilot test the feasibility and acceptability of a 12 week mHealth intervention to increase PA in metastatic breast cancer (MBC) patients using a two-arm randomized control trial (RCT). We will also examine the effects of the intervention on symptom burden, quality of life, and functional performance. Inactive MBC patients will be assigned to Fit2ThriveMB or education control. Participants assigned to the Fit2ThriveMB will receive the Fit2ThriveMB smartphone app, Fitbit, and coaching calls. Participants in the education control will be asked to download the app cancer.net from the American Society of Clinical Oncology, will receive educational materials and calls during the intervention period and the Fitbit following completion of 12 week assessments.

ELIGIBILITY:
Inclusion Criteria:

* Female; ≥18 years of age
* Diagnosed with metastatic breast cancer or locally advanced disease not amenable to surgical resection (Metastases to the auxiliary lymph nodes, and nowhere else in the body, do not qualify).
* Fluent in spoken and written English
* Own a smartphone
* Have access to the internet to complete assessments
* Self-report engaging in <150 minutes of moderate to vigorous PA per week.

Exclusion Criteria:

* Untreated brain metastases
* Uncontrolled cardiovascular disease or other major contraindications (i.e. non- ambulatory, severe cognitive or functional limitations) to PA participation
* Current enrollment in another dietary or PA trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be made available to other researchers in compliance with the NIH Data Sharing Policy. We welcome inquiries by investigators who are not associated with the study to review or analyze data that we have collected. All requests for data sharing will be handled by the PI, Dr. Phillips, in conjunction with co-investigators, on a case by case basis to ensure that the proposed work does not conflict with planned analyses; we will also establish that the proposed project has sufficient scientific merit before proceeding.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Phillips SM, Starikovsky J, Solk P, Desai R, Reading JM, Hasanaj K, Wang SD, Cullather E, Lee J, Song J, Spring B, Gradishar W. Feasibility and preliminary effects of the Fit2ThriveMB pilot physical activity promotion intervention on physical activity and patient reported outcomes in individuals with metastatic breast cancer. Breast Cancer Res Treat. 2024 Nov;208(2):391-403. doi: 10.1007/s10549-024-07432-5. Epub 2024 Jul 16. PMID 39014267
- [Derived] Phillips S, Solk P, Welch W, Auster-Gussman L, Lu M, Cullather E, Torre E, Whitaker M, Izenman E, La J, Lee J, Spring B, Gradishar W. A Technology-Based Physical Activity Intervention for Patients With Metastatic Breast Cancer (Fit2ThriveMB): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Apr 23;10(4):e24254. doi: 10.2196/24254. PMID 33890857

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fit2ThriveMB | Healthy Living Control
Started | 25 | 24
Completed | 24 | 24
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were included in baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fit2ThriveMB | Healthy Living Control | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (11.9) | 52.2 (29.7) | 54.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 21 | 21 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Number of Participants Randomized [Count of Participants; unit: Participants] | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Retained During the 12 Week Technology Supported Physical Activity Intervention Period
Description: Feasibility will be assessed via participant retention during the intervention period [(# of participants randomized- # of participants who drop out or are lost to follow-up)/ # randomized].
Time Frame: 12 weeks
Population: All participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
Participants | 24 | 24

2. Primary Outcome: Adherence to a 12 Week Technology Supported Physical Activity Intervention by Metastatic Breast Cancer Patients
Description: Adherence during the 12 week intervention will be monitored continuously using Fit2ThriveMB app. This measure the average percentage of days each participant in the Fit2ThriveMB intervention group wore the Fitbit.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days the Fitbit was worn.
Arm/Group | Fit2ThriveMB
Number analyzed (Participants) | 24
Percentage of days the Fitbit was worn. | 98.2 (2.5)

3. Primary Outcome: Acceptability of a 12 Week Technology Supported Physical Activity Intervention to Metastatic Breast Cancer Patients
Description: Acceptability will be measured via a process evaluation of perceptions of MBC patients' experiences with Fit2ThriveMB. Acceptability will be measured as the number of intervention participants who are satisfied/very satisfied with their overall study experience.
Time Frame: 12 weeks
Population: One participant did not complete the acceptability questionnaire at 12 weeks.
Measure: Number; unit: Participants
Arm/Group | Fit2ThriveMB
Number analyzed (Participants) | 23
Participants | 24

4. Secondary Outcome: Change in Physical Activity Minutes From Before to After a 12 Week Technology Supported Physical Activity Intervention in Metastatic Breast Cancer Patients
Description: Physical activity will be measured at baseline and at 12 weeks. The change between physical activity at baseline and 12-weeks will be assessed. The ActiGraph accelerometer will be used. At each time point, participants will wear the device for 7 consecutive days during all waking hours, except when bathing or swimming. Each valid minute of wear time will be classified according to intensity (counts/min) using commonly accepted cut-points: sedentary (<100), light activity (100-2019) and moderate/vigorous physical activity (≥2020).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
Minutes | -3.5 (56.6) | -18.7 (63.09)

5. Secondary Outcome: Change in Quality of Life From From Baseline to 12-weeks
Description: Quality of life will be measured at baseline and 12 weeks using the Functional Assessment of Cancer Therapy-Breast (FACT-B). Totals scores range from 0 to 148. Higher scores indicate better quality of life.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
score on a scale | 1.7 (1.9) | 2.0 (1.8)

6. Secondary Outcome: Change in Anxiety From Baseline to 12-weeks
Description: Anxiety will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Anxiety 8a health measure. T-scores range from 37.1 to 83.1. Higher scores indicate more anxiety. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
t-score on a scale | 0.8 (1.2) | 1.1 (1.2)

7. Secondary Outcome: Change in Depression From Baseline to 12-weeks
Description: Depression will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Depression 8a health measure. T-scores range from 38.2 to 81.3. Higher scores indicate more depression. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
t-score on a scale | 0.1 (1.3) | -0.05 (1.3)

8. Secondary Outcome: Change in Fatigue From Baseline to 12-weeks
Description: Fatigue will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue 8a health measure. T-scores range from 33.1 to 77.8 Higher scores indicate more fatigue. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
t-score on a scale | -2.7 (1.3) | 0.6 (1.3)

9. Secondary Outcome: Change in Pain Interference From Baseline to 12-weeks
Description: Pain Interference will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Pain Interference 8a health measure. T-scores range from 40.7 to 77.0 Higher scores indicate more pain interference.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
score on a scale | 3.2 (1.8) | -1.5 (1.8)

10. Secondary Outcome: Change in Physical Function From Baseline to 12-weeks
Description: Physical function will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-physical function 20a health measure. T-scores range from 32.7 to 62.7. Higher scores indicate better physical functioning. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
t-score on a scale | -0.1 (1.3) | 1.4 (1.3)

11. Secondary Outcome: Change in Sleep Disturbance From Baseline to 12-weeks
Description: Sleep disturbance will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-sleep disturbance 8a health measure. T-scores range from 30.5 to 77.5. Higher scores more sleep disturbance. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 25 | 24
t-score on a scale | -0.3 (0.8) | -0.2 (0.8)

12. Secondary Outcome: Change in Short Physical Performance Battery (SPPB) Scores From Baseline to 12 Weeks
Description: Participants will complete the Short Physical Performance Battery which includes assessments of gait speed, chair stands and standing balance that are combined to obtain a SPPB score. This test will be conducted at baseline and 12 weeks. SPPB scores range from 0 to 12. Higher scores mean better physical functioning.
Time Frame: Baseline and 12 weeks
Population: The SPPB was only conducted on a subset of participants due to disruptions in research related to the COVID-19 pandemic.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 12 | 11
score on a scale | .41 (.29) | -.55 (.37)

13. Secondary Outcome: Change in Arm Curl Test and Two-Minute Step Test From the Senior Fitness Test Measures Between Baseline and 12 Weeks
Description: The Senior Fitness Test measures physical function. The arm curl test assesses the number of times (repetitions) a 5lb hand-weight is curled in 30 seconds. The 2-minute step test evaluates the number of times (repetitions) the right knee reaches a distance half way between the iliac crest and patella during 2-minutes. Increased number of repetitions on both tests represents better physical function.
Time Frame: Baseline and 12 weeks
Population: The Senior Fitness Test was conducted on a subset of participants due to disruptions in research caused by the COVID-19 pandemic.
Measure: Mean (Standard Error); unit: Repetitions
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 12 | 11
Repetitions
  Arm Curl Test | 1.42 (0.96) | 2.91 (2.48)
  2-Minute Step Test | 12.92 (5.16) | 3.70 (4.87)

14. Secondary Outcome: Change in 6-minute Walk Test Distance Between Baseline and 12-weeks.
Description: Participants will complete a 6 minute walk test at baseline and 12 weeks. Distance is measured in meters. Increases in distance represent better performance.
Time Frame: Baseline and 12 weeks
Population: The 6-minute walk test was conducted on a subset of participants due to disruptions in research caused by the COVID-19 pandemic.
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 12 | 11
Meters | 19.42 (17.4) | 15.10 (5.50)

15. Secondary Outcome: Change in One Leg Stand Test and 8-foot-up-and go From the Senior Fitness Test Measures Between Baseline and 12 Weeks
Description: The Senior Fitness Test measures physical function. The one leg stand test assesses how long an individual can stand on each of their feet (right and left) in seconds up to 30-seconds. Increases in time on the one leg stand tests indicate better functioning. The 8-foot up and go test assesses how long it takes in seconds to stand from a chair, walk 8 feet around an object and return to sitting. Decreases in time indicate better functioning.
Time Frame: Baseline and 12 weeks
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Fit2ThriveMB | Healthy Living Control
Number analyzed (Participants) | 12 | 11
Seconds
  One Leg Stand: Right Leg | 1.48 (1.84) | -1.33 (2.71)
  One Leg Stand: Left Leg | 4.40 (2.64) | 1.87 (1.04)
  8-foot-up-and-go | -0.23 (0.26) | 0.29 (0.40)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 12 weeks.
Description: Participants were instructed to notify the study team immediately if they experienced any adverse events and were sent a survey every 4 weeks during the 12 week intervention to ask about any events that may have occurred over the past 4 weeks.
Arm/Group | Fit2ThriveMB | Healthy Living Control
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT04129346/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT04129346/ICF_001.pdf